CLINICAL TRIAL: NCT06850077
Title: Comparison of Prefrontal Hemodynamic Responses and Balance Control Differences Based on Head Posture and Task Difficulty in Cognitive-Balance Tasks
Status: Completed | Type: Observational
Sponsor: Sahmyook University (Other)
Responsible Party: Principal Investigator, Kim jeong eun, Principal Investigator (PI), Sahmyook University
Other Study IDs: SYU 2025-01-017-003
Record Dates: First submitted 2025-02-18; First posted 2025-02-27 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-09

CONDITIONS: Forward Head Posture; Normal Head Posture
Keywords: forward head posture; dual task; prefrontal cortex; cognition

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Forward head posture group: The experiment will be conducted for approximately 30 minutes. It will comprise cognitive tasks with three levels of difficulty and balance tasks, with task difficulty adjusted according to each participant's cognitive and balance abilities.
  During the experiment, changes in cerebral blood flow, cognitive performance, and balance ability will be assessed and analyzed.
  Interventions: Behavioral: Cognitive-Balance dual task
- Normal head posture group: The experiment will be conducted for approximately 30 minutes. It will comprise cognitive tasks with three levels of difficulty and balance tasks, with task difficulty adjusted according to each participant's cognitive and balance abilities.
  During the experiment, changes in cerebral blood flow, cognitive performance, and balance ability will be assessed and analyzed.
  Interventions: Behavioral: Cognitive-Balance dual task

INTERVENTIONS:
Behavioral: Cognitive-Balance dual task — The cognitive-balance dual task consists of three levels of difficulty and is performed simultaneously.
  The cognitive tasks include the N-back test, while the balance tasks consist of static balance tasks.

SUMMARY:
* Recent studies have shown that individuals with forward head posture (FHP) experience not only impaired balance control but also cognitive deficits.
* Using a balance-cognitive dual-task paradigm, this study aims to explore the relationship between balance ability and Prefrontal cortex(PFC) oxygenation levels(△HbO2) in individuals with FHP compared to those with normal head posture(NHP).
* By analyzing differences in frontal lobe activation based on task difficulty, this study is expected to provide practical data for designing balance training and cognitive-motor intervention programs tailored to individuals with FHP.

DETAILED DESCRIPTION:
- This study is a cross-sectional study aiming to investigate the differences in balance ability between individuals with forward head posture (FHP) and those with normal head posture (NHP), as well as the differences in frontal lobe oxygenation levels during a balance-cognitive dual task.

Study participants will be assigned to receive two groups: (a) Forward head posture (b) Normal head posture. Each group will perform three balance tasks while simultaneously completing three cognitive tasks. To determine the differences, the primary outcome will assess prefrontal cortex (PFC) hemodynamic response, and the secondary outcome will assess balance ability.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 20 to 39 years
* Classified as having Forward Head Posture (FHP) or Normal Head Posture (NHP) based on Craniovertebral Angle (CVA) measurement

Exclusion Criteria:

* Individuals with a history of spinal or musculoskeletal trauma or surgery
* Individuals who have reported recent neck or shoulder pain

Ages: 20 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants will be recruited from Samyook University(Seoul, South Korea) or local communities in Daegu or Seoul, South Korea. Recruitment will primarily target individuals who regularly engage in academic or sedentary activities. The study population will consist of individuals classified based on postural characteristics, specifically Forward Head Posture (FHP) or Normal Head Posture (NHP), assessed using craniovertebral angle (CVA) measurements. Recruitment will take place through campus advertisements, online postings, and word-of-mouth referrals.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2025-04-27 (Actual); Primary Completion 2025-10-20 (Actual); Study Completion 2025-10-20 (Actual)

PRIMARY OUTCOMES:
The degree of hemodynamic response in the prefrontal cortex (PFC) | From enrollment to 2 days
  Hemodynamic response changes in the prefrontal cortex (PFC) will be assessed by measuring variations in oxyhemoglobin (HbO) concentration using functional near-infrared spectroscopy (fNIRS). The study will compare HbO concentration changes between the control and experimental groups during cognitive-balance task performance.

SECONDARY OUTCOMES:
Balance performance | From enrollment to 2 days
  Static and dynamic balance performance will be assessed using the Good Balance system (Metitur, Finland). The assessment will be conducted on a triangular platform by measuring changes in the center of pressure (COP), regardless of foot position. The results will be reported as variations in COP displacement and velocity.
  Dynamic balance performance will be assessed using the Four Square Step Test (FSST). Participants will step in four quadrants formed by rods or tape arranged in a cross pattern. The time taken to complete the FSST will be recorded in seconds.

CONTACTS AND LOCATIONS:
Locations (1):
- Sahmyook university, Seoul, 노원구, South Korea

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 3 years after the publication of results